CLINICAL TRIAL: NCT03086655
Title: Tel-Me-Box: Validating and Testing a Novel, Low-cost, Real-time Monitoring Device With Hair Level Analysis Among Adherence-challenged Patients
Brief Title: Tel-Me-Box: Testing a New, Real-time Strategies for Monitoring HIV Medication Adherence in India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: R01MH109310 (NIH); R01MH109310 (NIH)
Record Dates: First submitted 2017-03-16; First posted 2017-03-22 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: HIV; Medication Adherence
Keywords: biological markers; monitoring device; wireless technology
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pillbox ('Tel-me-box') with reminder features (Experimental): Participants randomly assigned to the intervention reminder condition will choose from the reminders available and convey their preferences regarding when reminders should be sent for the tel-me-box device.
  Interventions: Behavioral: Tel-me-box with reminder features
- Pillbox ('Tel-me-box') without reminder features (Other): The control arm will include tel-me-box monitoring only. No reminder features will be included with the device.
  Interventions: Behavioral: Tel-me-box

INTERVENTIONS:
Behavioral: Tel-me-box with reminder features — Participants will meet with a study staff member to go over their daily routines, including their pill taking schedule, and to work out a plan for tailored reminders. The participant will choose from the reminders available and convey their preferences regarding when reminders should be sent for the TMB. Preferences will be stored in an online secure database. If requested by the participant, the reminder schedule and type of reminder can be reprogrammed by study staff via an online portal. When the reminder is reprogrammed the TMB receives a new configuration SMS to update the device reminder settings.
  Arms: Pillbox ('Tel-me-box') with reminder features
Behavioral: Tel-me-box — Participants receive tel-me-box device with no reminder features added.
  Arms: Pillbox ('Tel-me-box') without reminder features

SUMMARY:
Currently available methods to monitor antiretroviral (ARV) adherence to HIV treatment and prevention, such as self-report, pill counts, medication electronic monitoring system (MEMS), and devices which wirelessly monitor adherence in real-time, have multiple limitations, including over-reporting, inability to assess pill ingestion, and size/expense. Our multidisciplinary research team at the University of California, San Francisco (UCSF) and in India has designed a new adherence-monitoring device called "Tel-Me-Box" which is small, low-cost, rechargeable, inconspicuous, and could be programmed to deliver tailored real-time adherence reminders following additional hardware modifications. The aim of this study is to modify and validate this discreet Tel-Me-Box (TMB) adherence monitoring and reminder device against hair ARV concentrations as a pharmacologic measure of drug ingestion/adherence, a measure pioneered and validated by our team, with the expectation that this device and intermittent hair monitoring could have widespread utility for HIV and non-HIV adherence science, both in India and globally.

DETAILED DESCRIPTION:
Novel, validated methods to monitor adherence to HIV treatment in real time are urgently needed given the well-known limitations of self-reported adherence, pill counts, and MEMS caps. In order to be scalable and sustainable in both resource-rich and resource limited settings, such devices need to be low-cost and designed in a way that does not increase the risk of accidental HIV disclosure and subsequent stigma. Devices which both monitor adherence in real time and provide tailored reminders to patients for medication-taking have the potential to greatly improve adherence to HIV treatment as well as to treatment for other chronic diseases. Our Indo-US collaborative team has been conducting research on HIV stigma, ARV adherence patterns and barriers, treatment outcome, and drug resistance for over a decade. The study investigators have also pioneered the use of ARV concentrations in small hair samples to measure long-term ARV adherence in resource-rich and limited settings (RLS). In response to the need for novel adherence measures, our team has recently developed Tel-Me-Box, a small, low-cost adherence device that monitors adherence in real time, by transmitting a wireless signal to a server when opened. The investigators now propose to add hardware that will enable the server software to wirelessly program the device to activate tailored medication-taking reminders (via a beep, vibration, or LED light) after a period of inactivity. The device fits in a pocket, can hold 1-2 weeks' worth of medications, has a long battery life, simple charging capability, and has been found acceptable to Indian patients with adherence challenges in pilot studies. Since HIV stigma serves as a profound barrier to ARV adherence in many settings, including India, the small, inconspicuous nature of Tel-Me-Box, along with its ability to deliver tailored reminder features honors participants' privacy concerns. Since this electronic device monitoring cannot assess actual drug ingestion, validating it against a biological measure of adherence, such as ARV hair concentrations, is crucial.

This study includes a pilot randomized control trial (RCT) to examine acceptability and feasibility and to estimate the effect size of automated tailored real-time adherence reminders on hair ARV concentrations, device- monitored adherence, and viral load suppression in adherence-challenged patients.

The aim of this study is to validate TMB as an innovative tool to assess adherence and predict treatment outcomes, and demonstrate the feasibility of hair analyses in RLS. If successful, pilot data will be available on the efficacy of the Tel-Me-Box automated, tailored reminders for a future large scale RCT.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive
* Currently on antiretroviral therapy (ART)
* Speaks one of the local languages
* Able and willing to participate in the study, provide informed consent, contact information, and express a willingness to return for follow-up visits every three months for 12 months after baseline.
* Adherence-challenged per self-report, i.e. report of <90% ART adherence or >2 ART treatment interruptions of at least 2 days in the past 3 months

Exclusion Criteria:

* Unwilling or unable to participate in the study and/or return for follow-up appointments
* younger than 18 years old
* Not HIV-infected
* Not currently on ART
* Does not speak one of the local languages

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2021-08-13 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Ekstrand, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- St. John & Research Institute/St John & Medical College & Hospital, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Farmer KC. Methods for measuring and monitoring medication regimen adherence in clinical trials and clinical practice. Clin Ther. 1999 Jun;21(6):1074-90; discussion 1073. doi: 10.1016/S0149-2918(99)80026-5. PMID 10440628
- [Background] Chesney MA. The elusive gold standard. Future perspectives for HIV adherence assessment and intervention. J Acquir Immune Defic Syndr. 2006 Dec 1;43 Suppl 1:S149-55. doi: 10.1097/01.qai.0000243112.91293.26. PMID 17133199
- [Background] Berg KM, Arnsten JH. Practical and conceptual challenges in measuring antiretroviral adherence. J Acquir Immune Defic Syndr. 2006 Dec 1;43 Suppl 1(Suppl 1):S79-87. doi: 10.1097/01.qai.0000248337.97814.66. PMID 17133207
- [Background] Kripalani S, Yao X, Haynes RB. Interventions to enhance medication adherence in chronic medical conditions: a systematic review. Arch Intern Med. 2007 Mar 26;167(6):540-50. doi: 10.1001/archinte.167.6.540. PMID 17389285
- [Background] Nair BG, Newman SF, Peterson GN, Wu WY, Schwid HA. Feedback mechanisms including real-time electronic alerts to achieve near 100% timely prophylactic antibiotic administration in surgical cases. Anesth Analg. 2010 Nov;111(5):1293-300. doi: 10.1213/ANE.0b013e3181f46d89. Epub 2010 Sep 14. PMID 20841414
- [Background] Patel UB, Ni Q, Clayton C, Lam P, Parks J. An attempt to improve antipsychotic medication adherence by feedback of medication possession ratio scores to prescribers. Popul Health Manag. 2010 Oct;13(5):269-74. doi: 10.1089/pop.2009.0053. PMID 20879908
- [Background] Ruppar TM. Randomized pilot study of a behavioral feedback intervention to improve medication adherence in older adults with hypertension. J Cardiovasc Nurs. 2010 Nov-Dec;25(6):470-9. doi: 10.1097/JCN.0b013e3181d5f9c5. PMID 20856132
- [Background] Burgess SW, Sly PD, Devadason SG. Providing feedback on adherence increases use of preventive medication by asthmatic children. J Asthma. 2010 Mar;47(2):198-201. doi: 10.3109/02770900903483840. PMID 20170329
- [Background] Sabin LL, DeSilva MB, Hamer DH, Xu K, Zhang J, Li T, Wilson IB, Gill CJ. Using electronic drug monitor feedback to improve adherence to antiretroviral therapy among HIV-positive patients in China. AIDS Behav. 2010 Jun;14(3):580-9. doi: 10.1007/s10461-009-9615-1. PMID 19771504
- [Background] Cramer J, Rosenheck R, Kirk G, Krol W, Krystal J; VA Naltrexone Study Group 425. Medication compliance feedback and monitoring in a clinical trial: predictors and outcomes. Value Health. 2003 Sep-Oct;6(5):566-73. doi: 10.1046/j.1524-4733.2003.65269.x. PMID 14627063
- [Background] de Bruin M, Hospers HJ, van Breukelen GJ, Kok G, Koevoets WM, Prins JM. Electronic monitoring-based counseling to enhance adherence among HIV-infected patients: a randomized controlled trial. Health Psychol. 2010 Jul;29(4):421-8. doi: 10.1037/a0020335. PMID 20658830
- [Background] Vallabhaneni S, Chandy S, Heylen E, Ekstrand ML. Evaluation of WHO immunologic criteria for treatment failure: implications for detection of virologic failure, evolution of drug resistance and choice of second-line therapy in India. J Int AIDS Soc. 2013 Jun 3;16(1):18449. doi: 10.7448/IAS.16.1.18449. PMID 23735817
- [Background] Bachman Desilva M, Gifford AL, Keyi X, Li Z, Feng C, Brooks M, Harrold M, Yueying H, Gill CJ, Wubin X, Vian T, Haberer J, Bangsberg D, Sabin L. Feasibility and Acceptability of a Real-Time Adherence Device among HIV-Positive IDU Patients in China. AIDS Res Treat. 2013;2013:957862. doi: 10.1155/2013/957862. Epub 2013 Jul 16. PMID 23956851
- [Background] Vallabhaneni S, Chandy S, Heylen E, Ekstrand M. Reasons for and correlates of antiretroviral treatment interruptions in a cohort of patients from public and private clinics in southern India. AIDS Care. 2012;24(6):687-94. doi: 10.1080/09540121.2011.630370. Epub 2011 Nov 22. PMID 22107044
- [Background] Steward WT, Herek GM, Ramakrishna J, Bharat S, Chandy S, Wrubel J, Ekstrand ML. HIV-related stigma: adapting a theoretical framework for use in India. Soc Sci Med. 2008 Oct;67(8):1225-35. doi: 10.1016/j.socscimed.2008.05.032. Epub 2008 Jul 1. PMID 18599171
- [Background] Steward WT, Chandy S, Singh G, Panicker ST, Osmand TA, Heylen E, Ekstrand ML. Depression is not an inevitable outcome of disclosure avoidance: HIV stigma and mental health in a cohort of HIV-infected individuals from Southern India. Psychol Health Med. 2011 Jan;16(1):74-85. doi: 10.1080/13548506.2010.521568. PMID 21218366
- [Background] Steward WT, Bharat S, Ramakrishna J, Heylen E, Ekstrand ML. Stigma is associated with delays in seeking care among HIV-infected people in India. J Int Assoc Provid AIDS Care. 2013 Mar-Apr;12(2):103-9. doi: 10.1177/1545109711432315. Epub 2012 Jan 26. PMID 22282878
- [Background] Shet A, DeCosta A, Heylen E, Shastri S, Chandy S, Ekstrand M. High rates of adherence and treatment success in a public and public-private HIV clinic in India: potential benefits of standardized national care delivery systems. BMC Health Serv Res. 2011 Oct 17;11:277. doi: 10.1186/1472-6963-11-277. PMID 22004573
- [Background] Setia MS, Lindan C, Jerajani HR, Kumta S, Ekstrand M, Mathur M, Gogate A, Kavi AR, Anand V, Klausner JD. Men who have sex with men and transgenders in Mumbai, India: an emerging risk group for STIs and HIV. Indian J Dermatol Venereol Leprol. 2006 Nov-Dec;72(6):425-31. doi: 10.4103/0378-6323.29338. PMID 17179617
- [Background] Rodriguez DC, Krishnan AK, Kumarasamy N, Krishnan G, Solomon D, Johnson S, Vasudevan CK, Solomon R, Ekstrand ML. Two sides of the same story: alcohol use and HIV risk taking in South India. AIDS Behav. 2010 Aug;14 Suppl 1(Suppl 1):S136-46. doi: 10.1007/s10461-010-9722-z. PMID 20544382
- [Background] Nyamathi AM, William RR, Ganguly KK, Sinha S, Heravian A, Albarran CR, Thomas A, Greengold B, Ekstrand M, Ramakrishna P, Rao PR. Perceptions of Women Living with AIDS in Rural India Related to the Engagement of HIV-Trained Accredited Social Health Activists for Care and Support. J HIV AIDS Soc Serv. 2010 Oct;9(4):385-404. doi: 10.1080/15381501.2010.525474. PMID 21331322
- [Background] Nyamathi AM, Sinha S, Ganguly KK, William RR, Heravian A, Ramakrishnan P, Greengold B, Ekstrand M, Rao PV. Challenges experienced by rural women in India living with AIDS and implications for the delivery of HIV/AIDS care. Health Care Women Int. 2011 Apr;32(4):300-13. doi: 10.1080/07399332.2010.536282. PMID 21409663
- [Background] Navani-Vazirani S, Solomon D, Gopalakrishnan, Heylen E, Srikrishnan AK, Vasudevan CK, Ekstrand ML. Mobile phones and sex work in South India: the emerging role of mobile phones in condom use by female sex workers in two Indian states. Cult Health Sex. 2015;17(2):252-65. doi: 10.1080/13691058.2014.960002. Epub 2014 Oct 10. PMID 25301669

RESULTS

PARTICIPANT FLOW:
Period: Baseline Assessment
Arm/Group | Pillbox ('Tel-me-box') With Reminder Features | Pillbox ('Tel-me-box') Without Reminder Features
Started | 69 | 62
Completed | 69 | 62
Not Completed | 0 | 0
Period: 3 Month Follow-up Assessment
Arm/Group | Pillbox ('Tel-me-box') With Reminder Features | Pillbox ('Tel-me-box') Without Reminder Features
Started | 69 | 62
Completed | 62 | 58
Not Completed | 7 | 4
Not completed — Lost to Follow-up | 5 | 4
Not completed — Withdrawal by Subject | 2 | 0
Period: 6 Month Follow-up Assessment
Arm/Group | Pillbox ('Tel-me-box') With Reminder Features | Pillbox ('Tel-me-box') Without Reminder Features
Started | 67 (Number started = 67 = 69 randomized to this arm - 2 who withdrew at 3 mo follow-up. Study continued to try to reach those who were lost to follow-up in previous period.) | 62 (Number started = 62 because no subjects withdrew and study continued to try to reach those who were lost to follow-up in previous period.)
Completed | 58 | 55
Not Completed | 9 | 7
Not completed — Lost to Follow-up | 7 | 6
Not completed — Withdrawal by Subject | 2 | 1
Period: 9 Month Follow-up Assessment
Arm/Group | Pillbox ('Tel-me-box') With Reminder Features | Pillbox ('Tel-me-box') Without Reminder Features
Started | 65 (Number who started = 65 = 69 who started at baseline - 4 withdrawn in earlier periods) | 61 (Number started = 61 = 62 at baseline - 1 withdrawn at 6 mo.)
Completed | 56 | 57
Not Completed | 9 | 4
Not completed — Lost to Follow-up | 9 | 4
Period: 12 Month Follow-up = Final Assessment
Arm/Group | Pillbox ('Tel-me-box') With Reminder Features | Pillbox ('Tel-me-box') Without Reminder Features
Started | 65 (Number who started = 65 = 69 who started at baseline - 4 withdrawn in earlier periods) | 61 (Number started = 61 = 62 at baseline - 1 withdrawn at 6 mo.)
Completed | 58 | 57
Not Completed | 7 | 4
Not completed — Lost to Follow-up | 7 | 3
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pillbox ('Tel-me-box') With Reminder Features | Pillbox ('Tel-me-box') Without Reminder Features | Total
Number analyzed (Participants) | 69 | 62 | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (10.1) | 41.8 (9.6) | 39.4 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 26 | 61
  Male | 34 | 36 | 70
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 69 | 62 | 131
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  India | 69 | 62 | 131
Type of reminder feature (in intervention group only) [Count of Participants; unit: Participants]
  Buzzer | 34 | 0 | 34
  Light + vibration | 35 | 0 | 35
  None (only applicable to arm without reminder features) | 0 | 62 | 62

OUTCOME MEASURES:

1. Primary Outcome: Tel-me-box Adherence
Description: Number of days over past 30 days with at least one device-recorded pill box opening.
Time Frame: 30 days prior to each follow-up assessment (3, 6, 9 and 12 months post baseline).
Population: Overall number analyzed = number of participants enrolled at baseline. Numbers analyzed reported below reflect missing data due to loss to follow-up.
Measure: Median (Inter-Quartile Range); unit: days (out of 30)
Arm/Group | Pillbox ('Tel-me-box') With Reminder Features | Pillbox ('Tel-me-box') Without Reminder Features
Number analyzed (Participants) | 69 | 62
days (out of 30)
  No. days box opened (0-30) at 3 mo. follow-up: number analyzed (Participants) | 62 | 58
  No. days box opened (0-30) at 3 mo. follow-up | 10 [1 to 24] | 16.5 [2 to 25]
  No. days box opened (0-30) at 6 mo. follow-up: number analyzed (Participants) | 58 | 55
  No. days box opened (0-30) at 6 mo. follow-up | 1.5 [0 to 12] | 7 [0 to 17]
  No. days box opened (0-30) at 9 mo. follow-up: number analyzed (Participants) | 56 | 57
  No. days box opened (0-30) at 9 mo. follow-up | 0 [0 to 2.5] | 1 [0 to 13]
  No. days box opened (0-30) at 12 mo. follow-up: number analyzed (Participants) | 58 | 57
  No. days box opened (0-30) at 12 mo. follow-up | 0 [0 to 1] | 0 [0 to 8]
Statistical Analysis 1: Comparison: Pillbox ('Tel-me-box') With Reminder Features vs Pillbox ('Tel-me-box') Without Reminder Features; We used zero inflated negative binomial regression due to the count variable being overdispersed and containing a large number of 0. The analysis aggregated over multiple time points per participant. It simultaneously tests the odds of having 0 openings and the difference in the rate of openings between the 2 intervention groups. These 2 results are reported separately. Null hypothesis 1: the odds of having 0 openings is lower in intervention than control group; Test type: Superiority; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.90 to 1.93] — This is the 'inflation part' of the zero inflated negative binomial model. We used cluster robust standard errors due to the multiple observations over time being nested within participant. Result shows odds of intervention group relative to control
Statistical Analysis 2: Comparison: Pillbox ('Tel-me-box') With Reminder Features vs Pillbox ('Tel-me-box') Without Reminder Features; We used zero inflated negative binomial regression due to the count variable being overdispersed and containing many 0s. The analysis aggregated over multiple time points per participant. It simultaneously tests the odds of having 0 openings and the difference in the rate of openings between the 2 intervention groups. These 2 results are reported separately. Null hypothesis 2: the incidence rate ratio for # days with box opening is >1, i.e. more openings in intervention than control group; Test type: Superiority; incidence rate ratio (IRR) = 0.77, 95% CI 2-sided [0.61 to 0.98] — This is the negative binomial part of the model. We used cluster robust standard errors due to the multiple observations being nested within participant. Result shows intervention group had lower rate of openings relative to control

2. Primary Outcome: HIV Viral Load (VL)
Description: HIV viral load (number of copies/ml of blood), dichotomized as undetectable VL (= suppressed, meaning <50 copies/ml detected) vs. detectable (or unsuppressed, meaning >= 50 copies/ml detected)
Time Frame: Baseline, and 6 and 12 month follow-up
Population: Overall number analyzed = number of participants enrolled at baseline. Numbers analyzed reported below reflect missing data for VL due to failed lab tests or loss to follow-up.
Measure: Number; unit: participants
Arm/Group | Pillbox ('Tel-me-box') With Reminder Features | Pillbox ('Tel-me-box') Without Reminder Features
Number analyzed (Participants) | 69 | 62
participants
  Undetectable VL at Baseline: number analyzed (Participants) | 68 | 61
  Undetectable VL at Baseline | 37 | 34
  Undetectable VL at 6mo FU: number analyzed (Participants) | 58 | 55
  Undetectable VL at 6mo FU | 34 | 45
  Undetectable VL at 12 mo FU: number analyzed (Participants) | 58 | 56
  Undetectable VL at 12 mo FU | 34 | 44
Statistical Analysis 1: Comparison: Pillbox ('Tel-me-box') With Reminder Features vs Pillbox ('Tel-me-box') Without Reminder Features; statistical analyses is a GEE model with logit link function and binomial distribution with odds of undetectable VL as outcome and as predictors: intervention, time and time*intervention. We hypothesize that over time, the odds of undetectable VL will be higher for the intervention than the control group, which would be reflected in a significant interaction effect time*intervention. H0: no significant interaction effect time*intervention; Test type: Superiority; p = 0.08, Chi-squared; overall Wald chi2 (2 d.f.), simultaneously testing if parameters for both 6 mo. by intervention and 12 mo. by intervention are different from 0

3. Primary Outcome: Hair Concentrations of Anti-retroviral Medications (ARV), in ng/mg
Description: Hair concentrations of Efavirenz (EFV) or Dolutegravir (DTG) in ng/mg, and log transformed to improve normality of the distribution if necessary. The vast majority of participants were on an ARV regimen that included either EFV or DTG at the time of the study.
Time Frame: 12 month follow-up
Population: Of the 131 participants who started the pilot trial, 111 were interviewed at 12 mo. follow-up. Ten of these participants were on a regimen that did not include EFV or DTG, resulting in n=101 for analysis.
Measure: Mean (Standard Deviation); unit: log10 transformed concentration (ng/mg)
Arm/Group | Pillbox ('Tel-me-box') With Reminder Features | Pillbox ('Tel-me-box') Without Reminder Features
Number analyzed (Participants) | 48 | 53
log10 transformed concentration (ng/mg) | 0.12 (0.71) | 0.28 (0.64)
Statistical Analysis 1: Comparison: Pillbox ('Tel-me-box') With Reminder Features vs Pillbox ('Tel-me-box') Without Reminder Features; Test type: Superiority; p < 0.05, t-test, 2 sided — a priori threshold for statistical significance was p=0.05; (equal variances assumed); Mean Difference (Net) = 0.16, 95% CI 2-sided [-0.11 to 0.43], Standard Error of Mean 0.13 — Difference = control group - treatment group

4. Secondary Outcome: Self-reported Adherence in the Past Month
Description: Participant self-report measured using the visual analogue scale to assess percent of pills taken in the past month, further dichotomized into optimal (100%) vs. suboptimal adherence (<100%)
Time Frame: 30 days prior to baseline and 3, 6, 9, and 12 month follow-up
Population: Overall number of participants = number enrolled at baseline. At follow-up waves the number analyzed is lower due to loss to follow-up.
Measure: Number; unit: participants
Arm/Group | Pillbox ('Tel-me-box') With Reminder Features | Pillbox ('Tel-me-box') Without Reminder Features
Number analyzed (Participants) | 69 | 62
participants
  Optimally adherent at baseline | 4 | 5
  Optimally adherent at 3 month follow up: number analyzed (Participants) | 62 | 58
  Optimally adherent at 3 month follow up | 49 | 37
  Optimally adherent at 6 month follow up: number analyzed (Participants) | 58 | 55
  Optimally adherent at 6 month follow up | 44 | 35
  Optimally adherent at 9 month follow up: number analyzed (Participants) | 56 | 57
  Optimally adherent at 9 month follow up | 45 | 40
  Optimally adherent at 12 month follow up: number analyzed (Participants) | 58 | 57
  Optimally adherent at 12 month follow up | 45 | 50
Statistical Analysis 1: Comparison: Pillbox ('Tel-me-box') With Reminder Features vs Pillbox ('Tel-me-box') Without Reminder Features; statistical analyses is a GEE model with logit link function and binomial distribution with odds of optimal adherence as outcome and as predictors: intervention, time and time*intervention. We hypothesize that over time, the odds of optimal adherence will be higher for the intervention than the control group, which would be reflected in a significant interaction effect time*intervention. H0: no significant interaction effect time*intervention; Test type: Superiority; p = 0.08, Chi-squared; overall Wald chi2 (4 d.f.), simultaneously testing if parameters for all follow-ups by intervention are different from 0

5. Post Hoc Outcome: Presence of Tel-me-box Adherence Data (>0) in Past 30 Days
Description: The number of participants for whom at least 1 pill box opening was registered in the 30 days before an assessment
Time Frame: 30 days prior to assessment at 3, 6, 9, and 12 mo follow-up
Measure: Number; unit: participants
Arm/Group | Pillbox ('Tel-me-box') With Reminder Features | Pillbox ('Tel-me-box') Without Reminder Features
Number analyzed (Participants) | 69 | 62
participants
  any box use data at 3 mo FU | 47 | 48
  any box use data at 6 mo FU | 38 | 41
  any box use data at 9 mo FU | 26 | 31
  any box use data at 12 mo FU | 16 | 22

ADVERSE EVENTS:
Time Frame: 1 year, i.e. between baseline and the final follow-up 12 months later
Arm/Group | Pillbox ('Tel-me-box') With Reminder Features | Pillbox ('Tel-me-box') Without Reminder Features
All-Cause Mortality (participants affected / at risk) | 0/69 | 1/62
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/62
Other Adverse Events (participants affected / at risk) | 0/69 | 0/62

LIMITATIONS AND CAVEATS:
This was a pilot RCT to determine the feasibility and acceptability of the intervention, and a preliminary estimate of its potential efficacy of adding reminder features to the study pillbox. It was NOT fully powered to test differences in adherence between those participants who did and those who did not have a reminder feature of their choice included in their Tel-me-box pill dispenser.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-07-02): https://cdn.clinicaltrials.gov/large-docs/55/NCT03086655/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-22): https://cdn.clinicaltrials.gov/large-docs/55/NCT03086655/SAP_001.pdf